CLINICAL TRIAL: NCT05459012
Title: Patient Education: Asthma and Pregnancy
Brief Title: Patient Education in Pregnant Women With Asthma
Acronym: TAPAGE
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO22079*
Record Dates: First submitted 2022-07-08; First posted 2022-07-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women with asthma
  Interventions: Other: follow-up

INTERVENTIONS:
Other: follow-up — Questionnaire of Quality of life

SUMMARY:
Pregnancy may impact treatment adherence in women with asthma. This is a major risk factor for asthma exacerbation, which may have an important impact for both women and the babies. This study aims to evaluate the impact of a targeted patient education action tailored for pregnant women with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women with asthma

Exclusion Criteria:

* women not able to speak and/or read French language
* women protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with asthma
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change from Asthma quality of life between two periods : before intervention and 3 month after the intervention | before and 3 month after the intervention
  The physician gives Asthma quality of life questionnaire (AQLQ) before intervention and 3 month after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided